CLINICAL TRIAL: NCT00782795
Title: Phase II Study of Chronic Pancreatitis and the Effect of Pioglitazone on Endocrine Function, Exocrine Function & Structure, Pain & Life Quality
Brief Title: Chronic Pancreatitis. Effect of Pioglitazone on Endocrine Function, Exocrine Function & Structure, Pain & Life Quality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew DiMagno, MD, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-PENQEX-1R21AA017271; R21AA017271 (NIH); 1R21AA017271-01A1 (NIH)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pancreatitis; Insulin Resistance; Normal or Mildly Abnormal Stool Fat Levels
Keywords: Chronic pancreatitis; Insulin resistance
MeSH Terms: conditions — Pancreatitis, Chronic; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): 30 mg pioglitazone (Actos) tablet taken once daily for 48 weeks.
  Interventions: Drug: Pioglitazone
- sugar pill (placebo) (Placebo Comparator): 1 sugar pill (placebo) taken once daily for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Participants randomized to pioglitazone receive 30 mg taken once daily for 48 weeks.
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo
  Arms: sugar pill (placebo)

SUMMARY:
The purpose of this study is to determine if study drug (Pioglitazone) treatment will improve pre-diabetes (insulin resistance) or ealy diabetes and improve clinical symptoms (pain) or laboratory evidence of chronic pancreatitis.

The goal of the investigators is to gather information from this study to help gain understanding of a potential therapy for chronic pancreatitis.

DETAILED DESCRIPTION:
The pancreas is a digestive organ that secretes insulin (and other hormones) into the blood for regulating blood sugar (glucose) and digestive enzymes into the intestine for digesting and absorbing nutrients consumed in meals. Chronic pancreatitis is a progressive clinical disease of the pancreas, associated with swelling (inflammation), scarring (fibrosis) and loss of normal functioning tissue. Patients develop diabetes mellitus (elevated blood sugar), malabsorption of nutrients, weight loss and pain. Presently chronic pancreatitis is considered an irreversible condition because the mechanisms responsible for chronic pancreatitis are poorly understood and no therapy is proven. However, recent studies provide important clues that oral medications (Thiazolidinediones) used to treat diabetes mellitus might improve or reverse features of chronic pancreatitis, including elevated sugar or diabetes, reduced secretion of digestive enzymes, and pancreatic swelling and scarring.

Note: Takeda Pharmaceuticals North America (TPNA) provided pioglitazone and placebo pills with identically appearance until June 28, 2010, approximately the middle of the study.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistance or mild diabetes mellitus
* Symptoms of abdominal pain
* Xray test showing damage to the pancreas
* Normal or mildly abnormal stool fat levels

Exclusion Criteria:

* Mentally disabled patients
* Women who are planning pregnancy, pregnant or lactating/nursing
* Chronic pancreatitis is due to other specific conditions

  * Autosomal dominant pancreatitis
  * Classic cystic fibrosis with lung involvement
  * Autoimmune pancreatitis
  * Pancreatic cancer
  * Biliary obstruction (non-pancreatic cause)
  * Abdominal trauma
  * Hypercalcemia
  * Hypertriglyceridemia
* Surgical resection of the head of the pancreas
* Alcohol consumption within prior 2 months
* Specific medical conditions

  * Gastric surgery
  * Celiac sprue
  * Crohns disease
  * Heart failure
  * Kidney failure
  * Cirrhosis or liver disease
  * Osteoporosis
  * Blood clotting disorder
  * Visual problems
  * Low albumin
  * Low BMI
* Specific medications *Diabetes drug treatment is allowed except for short-acting insulin, long-acting insule more than 15 units daily, pioglitazone, rosiglitazone, orlistat, acarbose, miglitol or voglibose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew DiMagno, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 screen fails did not go on to randomization
Groups:
- Pioglitazone: 30 mg pioglitazone (Actos) tablet taken once daily for 48 weeks.
  Pioglitazone: Participants will be randomized to either pioglitazone or placebo. The dosing is 30 mg taken once daily for 48 weeks.
- Sugar Pill (Placebo): 1 sugar pill (placebo) taken once daily for 48 weeks.
  Pioglitazone: Participants will be randomized to either pioglitazone or placebo. The dosing is 30 mg taken once daily for 48 weeks.
Period: Overall Study
Arm/Group | Pioglitazone | Sugar Pill (Placebo)
Started | 17 | 8
6 Weeks (1st Apptment) | 16 | 7
24 Week Appointment | 16 | 7
Completed | 16 | 6
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.35 (7.61) | 48.37 (9.83) | 51.08 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Glucose Tolerance at 24 Weeks
Description: 1. Normal = normal plasma glucose and normal glucose tolerance (OGTT).
  2. Impaired category includes all non-diabetic participants with either a) Impaired fasting glucose = fasting plasma glucose >110 mg/dl and <126 mg/dl; or b) Impaired glucose intolerance = 2-hour plasma glucose (OGTT) >140 mg/dl and <200 mg/dl.
  3. Diabetes = fasting plasma glucose >126 mg/dl 2-hour (OGTT) plasma glucose >200 mg/dl.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
Participants
  Diabetes | 2 | 4
  Impaired Glucose Tolerance | 3 | 4
  Normal | 2 | 8

2. Primary Outcome: Glucose Tolerance at 48 Weeks
Description: as for outcome 1
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
Participants
  Diabetes | 2 | 5
  Impaired Glucose Tolerance | 2 | 5
  Normal | 2 | 6

3. Primary Outcome: Insulin Sensitivity Index for Glycemia at 24 Weeks
Description: Insulin Sensitivity = Index for Glycemia (ISI gly) = 2 / ([INSp x GLYp] + 1).
  GLYp = Glycemic 0-2 hr area = sum of normalized (based on institutional values) 0 & 2 hr glucose.
  INSp = Insulinemic 0-2 hr area = sum of normalized (based on institutional values) 0 & 2 hr insulin.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: numeric index
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
numeric index | 0.26 (0.11) | 0.35 (0.20)

4. Primary Outcome: Insulin Sensitivity Index for Glycemia at 48 Weeks.
Description: as for outcome 3
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: numeric index
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
numeric index | 0.21 (0.13) | 0.36 (0.18)

5. Secondary Outcome: Beta-cell Function
Description: Homeostasis model assessment (HOMA 2) values generated using calculator at https://www.dtu.ox.ac.uk/homacalculator/
Time Frame: 24, 48 weeks
Population: 1 participant on the placebo side was no longer participating at 48 weeks
Measure: Mean (Standard Deviation); unit: Beta-cell function (%)
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
Beta-cell function (%)
  week 24 | 110.51 (31.59) | 120.59 (48.78)
  week 48: number analyzed (Participants) | 6 | 16
  week 48 | 121.60 (61.53) | 120.68 (44.39)

6. Secondary Outcome: Insulin Resistance at 24 and 48 Weeks
Description: Homeostasis model assessment (HOMA 2) values generated using calculator at https://www.dtu.ox.ac.uk/homacalculator/
Time Frame: 24, 48 weeks
Population: 1 participant on the placebo side was no longer participating at 48 weeks
Measure: Mean (Standard Deviation); unit: HOMA2-IR
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
HOMA2-IR
  24 weeks | 2.56 (1.29) | 2.27 (1.00)
  48 weeks: number analyzed (Participants) | 6 | 16
  48 weeks | 2.32 (0.85) | 2.42 (1.31)

7. Secondary Outcome: Pancreas Ultrasound Appearance
Description: Mean score on a scale of 0 - 10: count of positive Endoscopic Ultrasound(EUS) features:
  Parenchymal Features - Only Body and Tail
  1. Calcification (>3 hyperechoic foci >2 mm length & width with shadowing)
  2. Lobularity (>3 well-circumscribed, >5mm structures)
  3. Hyperechoic stranding (>3 hyperechoic lines >3mm in length, seen in > 2 different directions with respect to the imaged plane Parenchymal Features - Head, Body and Tail
  4. Cyst (>2 mm diameter anechoic round or oval structure)
  5. Hyperechoic foci (>3 reflectors, >3 mm long & wide, no shadowing) Ductal Features - Only Body and Tail
  6. Side Branch Dilation (>3 tubular, anechoic, >1 mm structures,Main pancreatic duct (MPD) connects)
  7. Irregular MPD contour (uneven and ectatic in its course)
  8. Hyperechoic MPD margin (hyperechoic in >50% of MPD)
  9. Dilation MPD (>3.5 mm body, >1.5 mm tail*) Ductal Features - Head, Body and Tail
  10. MPD calculi (hyperechoic foci with shadowing contained within MPD)
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
units on a scale | 4.5 [4 to 5] | 4.91 [3.5 to 6]

8. Secondary Outcome: Quality of Life
Description: The SF36 (Short Form with 36 questions) QoL scoring system has 36 questions, comprising two main dimensions (Physical Health and Mental Health), further divided by 8 independent scales (Physical functioning, Role-Physical, Bodily pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health). The scales for general health and mental health overlap components of both the two main dimensions (Physical Health and Mental Health). The scales, including the total score and dimensions are scored as a number between 0 and 100, where 0 represents lower limits of functioning and 100 is best functioning possible. Data reported is the average total score.
Time Frame: 24, 48 weeks
Population: The 24 week data has two participants' data missing from each arm because it was not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
units on a scale
  week 24: number analyzed (Participants) | 5 | 14
  week 24 | 67.74 (29.13) | 70.06 (18.86)
  week 48 | 66.0 (26.33) | 64.71 (23.54)

9. Secondary Outcome: Number and Percentage of Participants With Steatorrhea
Description: Participants were counted as having steatorrhea if they had either a) positive qualitative fecal fat; or b) 72 hour quantitative fecal fat result with >7g fat in stool in 24hours
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
Participants | 1 | 5

10. Secondary Outcome: Pain
Description: Pain is reported as the mean of four Visual analogue scales, ranging from 0 points (no pain) to 100 points (severe pain)
  1. What is your pain right now?
  2. What is your typical or average pain in the last 12 weeks?
  3. What is your pain level at its best in the last 12 weeks (how close to "0" does your pain get at its best)?
  4. What is your pain level at its worst in the last 12 weeks (how close to "0" does your pain get at its worst)?
Time Frame: 12, 24, 36, 48 and 60 weeks
Population: Some participant data is missing from some weeks, due to incomplete forms in certain instances.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
units on a scale
  week 12: number analyzed (Participants) | 6 | 16
  week 12 | 19.38 (21.46) | 23.03 (25.16)
  week 24: number analyzed (Participants) | 7 | 15
  week 24 | 26.32 (28.84) | 18.92 (22.71)
  week 36: number analyzed (Participants) | 6 | 15
  week 36 | 22.88 (21.97) | 23.55 (23.29)
  week 48: number analyzed (Participants) | 6 | 16
  week 48 | 25.42 (26.52) | 27.50 (27.88)
  week 60: number analyzed (Participants) | 5 | 16
  week 60 | 13.15 (16.08) | 26.11 (24.61)

11. Secondary Outcome: Body Mass Index (BMI)
Description: standard BMI defined as mass in kilograms divided by height in meters squared
Time Frame: 12, 24, 36, 48 and 60 weeks
Population: Some participant data is missing from some weeks, due to incomplete forms in certain instances.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 6 | 16
kg/m^2
  12 weeks | 28.02 (5.73) | 28.64 (6.88)
  24 weeks: number analyzed (Participants) | 5 | 15
  24 weeks | 25.56 (4.46) | 29.49 (6.36)
  36 weeks: number analyzed (Participants) | 6 | 14
  36 weeks | 28.55 (5.92) | 27.46 (6.01)
  48 weeks | 28.26 (6.36) | 28.75 (6.92)
  60 weeks: number analyzed (Participants) | 3 | 14
  60 weeks | 29.20 (4.36) | 27.94 (6.77)

12. Secondary Outcome: Hospitalizations
Description: Mean number of hospitalizations within the prior 12 weeks
Time Frame: 12, 24, 36, 48 and 60 weeks
Population: Some participant data is missing from some weeks, due to incomplete forms in certain instances.
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
hospitalizations
  week 12: number analyzed (Participants) | 6 | 16
  week 12 | 0 (0) | 0.06 (0.25)
  week 24 | 0.43 (1.13) | 0.06 (0.25)
  week 36: number analyzed (Participants) | 5 | 15
  week 36 | 0.20 (0.45) | 0.07 (0.26)
  week 48: number analyzed (Participants) | 6 | 16
  week 48 | 0 (0) | 0.12 (0.34)
  week 60: number analyzed (Participants) | 5 | 16
  week 60 | 0 (0) | 0.06 (0.25)

13. Secondary Outcome: Missed Work
Description: Mean days of missed work reported by participants in response to question asking about missed work since the last visit (12 weeks)
Time Frame: 12, 24, 36, 48, 60 weeks
Population: Some participant data is missing from some weeks, due to incomplete forms in certain instances.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
days
  week 12: number analyzed (Participants) | 6 | 16
  week 12 | 0.50 (1.20) | 0 (0)
  week 24 | 0.71 (1.89) | 0.75 (2.52)
  week 36: number analyzed (Participants) | 5 | 15
  week 36 | 0.20 (0.45) | 0.47 (1.36)
  week 48: number analyzed (Participants) | 6 | 16
  week 48 | 0 (0) | 0.5 (1.75)
  week 60 | 0 (0) | 0.25 (1)

14. Secondary Outcome: Insulin Sensitivity (%S)
Description: Homeostasis model assessment (HOMA 2) values generated using calculator at https://www.dtu.ox.ac.uk/homacalculator/;
Time Frame: 24 and 48 weeks
Population: 1 participant on the placebo side was no longer participating at 48 weeks
Measure: Mean (Standard Deviation); unit: insulin sensitivity (%)
Arm/Group | Sugar Pill (Placebo) | Pioglitazone
Number analyzed (Participants) | 7 | 16
insulin sensitivity (%)
  24 weeks | 45.39 (17.26) | 51.83 (20.42)
  48 weeks: number analyzed (Participants) | 6 | 16
  48 weeks | 48.12 (17.21) | 46.18 (26.86)

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: All adverse events that participants raised to study team as such, all of which were reported on to the IRB, are shown below.
Arm/Group | Pioglitazone | Sugar Pill (Placebo)
Serious Adverse Events (participants affected / at risk) | 4/17 | 2/8
Other Adverse Events (participants affected / at risk) | 0/17 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=17) | Sugar Pill (Placebo) (N=8)
chronic vertigo exacerbation (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 (8) | 1 (3)
Hyperglycemia (Endocrine disorders) | 0 | 1
Trauma to head (Nervous system disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
non-specific neck swelling (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes